CLINICAL TRIAL: NCT06517121
Title: Personalised Transcranial Direct Current Stimulation to Reduce Daily Loneliness in People With Subthreshold Depression
Brief Title: tDCS in People With Subthreshold Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: The University of Hong Kong (Other); Chinese University of Hong Kong (Other); Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, WONG Man Lok Nichol, Assistant Professor, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-2024-0048
Record Dates: First submitted 2024-07-11; First posted 2024-07-24 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Subthreshold Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalised tDCS group (Experimental): Participants who are assigned to the personalised group will receive anodal tDCS over a individualized stimulation site.
  Interventions: Device: Personalized Experimental Transcranial Direct Current Stimulation (tDCS)
- Conventional tDCS group (Experimental): Participants who are assigned to the Conventional group will receive anodal tDCS over F3.
  Interventions: Device: Conventional Experimental Transcranial Direct Current Stimulation (tDCS)
- Sham control group (Sham Comparator): Participants who are assigned to the Conventional group will receive sham tDCS. The active stimulation will be delivered for the first 30 seconds only.
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Personalized Experimental Transcranial Direct Current Stimulation (tDCS) — This study will deliver tDCS sessions for a maximum of ten sessions in two weeks' time. Participants will receive 20 minutes of active stimulation with a 2mA intensity over personalized brain regions based on the particular neural correlates of socio-affective processing.
  Arms: Personalised tDCS group
Device: Sham Transcranial Direct Current Stimulation (tDCS) — This study will deliver tDCS sessions for a maximum of ten sessions in two weeks' time. Participants assigned to the sham control group will only receive 30 seconds of active stimulation.
  Arms: Sham control group
Device: Conventional Experimental Transcranial Direct Current Stimulation (tDCS) — This study will deliver tDCS sessions for a maximum of ten sessions in two weeks' time. Participants will receive 20 minutes of active stimulation with a 2mA intensity with anode placed over F3.
  Arms: Conventional tDCS group

SUMMARY:
This study evaluates the effects of multi-session transcranial direct current stimulation on loneliness, mood and depressiveness in people with subthreshold depression.

DETAILED DESCRIPTION:
Depression-prone individuals will be invited and allocated to three groups, either the personalised transcranial direct current stimulation (tDCS) group, the conventional tDCS group, or the sham control group. After screening and at baseline prior to the tDCS sessions, participants will complete tests and questionnaires on depression symptoms, loneliness and mood. Eligible participants will also be invited to receive functional magnetic resonance imaging (MRI) in a 3-Tesla MRI scanner. There will be a maximum of 10 sessions to be completed after the screening and baseline measures. For both personalised tDCS group and the conventional tDCS group, tDCS with 2 milliampere (mA) intensity will be delivered for 20 minutes in each session. For sham control group, the protocol will be similar, except that the stimulation only happens in the first 30 seconds in each session. Especially for participants allocated to the personalised tDCS group, the stimulation site for each individual in this group may vary, depending on their brain activations and connectivity. The anodal stimulation sites for participants allocated to the conventional tDCS group and the sham control group will be F3 within the left DLPFC. Immediately after and also 3-months after completing all the tDCS sessions, participants will be invited to complete again tests and questionnaires on depressive symptoms in addition to loneliness and mood. Eligible participants will also be invited to receive functional MRI scanning in the 3T MRI scanner again. Participants will also be prompted to self-report daily their loneliness and mood levels throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* No histories of learning impairment, major psychiatric disorders including Major Depressive Disorder or neurological disorders
* At least primary school education
* Subthreshold depression

Exclusion Criteria:

* On medication or treatments within 2 weeks prior to the beginning of the study that would affect the individual's brain, cognitive and affective functions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Changes in self-reported loneliness | From baseline to after the last tDCS session; from baseline to 3 months after the last tDCS session
  Loneliness is assessed based on the University of California, Los Angeles (UCLA) loneliness scale and single item, in which higher scores indicate greater degrees of loneliness.

SECONDARY OUTCOMES:
Changes in depressive symptoms | From baseline to after the last tDCS session; from baseline to 3 months after the last tDCS session
  Depressive symptoms are assessed based on the Hospital Anxiety and Depression Scale, a 14-item scale assessing severity of depressive and anxiety symptom (score range 0 - 21 for both subscale), with a higher scores indicating higher severity
Changes in anxiety symptoms | From baseline to after the last tDCS session; from baseline to 3 months after the last tDCS session
  Anxiety symptoms are assessed based on the Hospital Anxiety and Depression Scale, a 14-item scale assessing severity of depressive and anxiety symptom (score range 0 - 21 for both subscale), with a higher scores indicating higher severity
Changes in self-reported mood | From baseline to after the last tDCS session; from baseline to 3 months after the last tDCS session
  Mood is assessed based on the Chinese Affect Scale, a 20-item 5-point Likert scale where participants rate the degree to which they currently feel the listed affects (scoring for each item: 0 = no at all; 4 = very).
Changes in brain activation and connectivity | From baseline to after the last tDCS session; from baseline to 3 months after the last tDCS session
  Neural activities and connectivity in Ventral Attention Network, Frontoparietal Network, and Default Mode Network are assessed by functional MRI

CONTACTS AND LOCATIONS:
Overall Officials: Nichol ML Wong, PhD, Principal Investigator — Education University of Hong Kong
Locations (1):
- The Education University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No